CLINICAL TRIAL: NCT00351169
Title: A Multi-Centre, Double-Blind, Randomised, Parallel Group, Placebo- Controlled and Active Controlled Phase III Study of the Efficacy and Safety of Quetiapine Fumarate Sustained Release (Seroquel SRTM) as Mono- Therapy in the Treatment of Adult Patients With Major Depressive Disorder
Brief Title: Efficacy of Seroquel SR in Combination With an Antidepressant in Treatment of Major Depressive Disorder
Acronym: AMBER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1448C00004; AMBER; EUDRACT No: 2005-005052-40
Record Dates: First submitted 2006-07-11; First posted 2006-07-12 (Estimated); Last update posted 2008-12-22 (Estimated); Status verified 2007-12

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; MDD
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram

INTERVENTIONS:
Drug: Quetiapine SR
Drug: Escitalopram

SUMMARY:
To evaluate the efficacy and safety of quetiapine fumarate sustained release (Seroquel SR) in the treatment of Major Depressive Disorder.

PLEASE NOTE: Seroquel SR and Seroquel XR refer to the same formulation. The SR designation was changed to XR after consultation with FDA.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 65 years
* A documented diagnosis of major depressive disorder

Exclusion Criteria:

* Patients with a DSM IV Axis I disorder other than MDD within 6 months of enrolment
* Patients with a diagnosis of DSM IV Axis II disorder which has a major impact on the patient's current psychiatric status
* Patients whose current episode of depression exceeds 12 months or is less than 4 weeks prior to enrolment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2006-05; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of quetiapine SR compared with placebo in the treatment of patients with major depressive disorder (MDD) as assessed by change from randomisation to week 8 score in the MADRS total score.

SECONDARY OUTCOMES:
If quetiapine SR improves health-related quality of life of patients with MDD, compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Willie Earley, MD, Study Director — AstraZeneca
Locations (42):
- Canada (14):
  - Research Site, Edmonton, Alberta
  - Research Site, Kelowna, British Columbia
  - Research Site, Penticton, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Sydney, Nova Scotia
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Oakville, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Gatineau, Quebec
  - Research Site, Montreal, Quebec
- China (5):
  - Research Site, Beijing
  - Research Site, HA Erbing
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Wuhan
- Finland (4):
  - Research Site, Helsinki
  - Research Site, Oulu
  - Research Site, Tampere
  - Research Site, Turku
- Malaysia (3):
  - Research Site, Johor Bahru
  - Research Site, Perak
  - Research Site, Petaling Jaya
- Mexico (3):
  - Research Site, Aguascalientes
  - Research Site, Distrito Federal
  - Research Site, Guadalajara
- Philippines (4):
  - Research Site, Cebu City
  - Research Site, Davao City
  - Research Site, Mandaluyong
  - Research Site, Manila
- South Africa (5):
  - Research Site, Benoni
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, Johannesburg
  - Research Site, Krugersdorp
- Research Site, Seoul, South Korea
- Spain (3):
  - Research Site, Langreo
  - Research Site, Vigo
  - Research Site, Zamora

REFERENCES:
- [Derived] McIntyre RS, Gorwood P, Thase ME, Liss C, Desai D, Chen J, Bauer M. Early Symptom Improvement as a Predictor of Response to Extended Release Quetiapine in Major Depressive Disorder. J Clin Psychopharmacol. 2015 Dec;35(6):706-10. doi: 10.1097/JCP.0000000000000416. PMID 26474010
- [Derived] Weisler R, Montgomery SA, Earley WR, Szamosi J, Eriksson H. Extended release quetiapine fumarate in patients with major depressive disorder: suicidality data from acute and maintenance studies. J Clin Psychiatry. 2014 May;75(5):520-7. doi: 10.4088/JCP.13m08624. PMID 24816198
- [Derived] Weisler R, McIntyre RS. The role of extended-release quetiapine fumarate monotherapy in the treatment of patients with major depressive disorder. Expert Rev Neurother. 2013 Nov;13(11):1161-82. doi: 10.1586/14737175.2013.846520. PMID 24175720
- [Derived] Clayton AH, Locklear JC, Svedsater H, McIntyre RS. Sexual functioning in patients with major depressive disorder in randomized placebo-controlled studies of extended release quetiapine fumarate. CNS Spectr. 2014 Apr;19(2):182-96. doi: 10.1017/S1092852913000631. Epub 2013 Sep 25. PMID 24067192
- [Derived] Trivedi MH, Bandelow B, Demyttenaere K, Papakostas GI, Szamosi J, Earley W, Eriksson H. Evaluation of the effects of extended release quetiapine fumarate monotherapy on sleep disturbance in patients with major depressive disorder: a pooled analysis of four randomized acute studies. Int J Neuropsychopharmacol. 2013 Sep;16(8):1733-44. doi: 10.1017/S146114571300028X. Epub 2013 May 14. PMID 23673347
- [Derived] Thase ME, Montgomery S, Papakostas GI, Bauer M, Trivedi MH, Svedsater H, Locklear JC, Gustafsson U, Datto C, Eriksson H. Quetiapine XR monotherapy in major depressive disorder: a pooled analysis to assess the influence of baseline severity on efficacy. Int Clin Psychopharmacol. 2013 May;28(3):113-20. doi: 10.1097/YIC.0b013e32835fb971. PMID 23485955